CLINICAL TRIAL: NCT00500955
Title: A Study to Evaluate the Efficacy of Rosiglitazone (BRL-049653) on Reduction of Microalbuminuria in Subjects With Type 2 Diabetes Mellitus
Brief Title: Rosiglitazone on Microalbuminuria in Type 2 Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRL-49653/137
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: microalbuminuria,; Type 2 Diabetes; rosiglitazone,
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
Following a 4-week single-blind placebo run-in period, eligible subjects were randomized in a 1:1 ratio to receive 32 weeks of double-blind study medication: Rosiglitazone (starting dose 4mg od) or Glyburide (starting dose 5mg od), both in combination with open-label Metformin > or = (1g/day). Subjects were stratified for use of ACEI, nondihydropyridine calcium channel blockers (NDP CCB), or angiotensin II receptor blockers (ARB) to provide equal representation of these subjects in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 40-80 with T2DM and Microalbuminuria previously treated by diet and exercise alone, a single oral antidiabetic agent, or combination oral antidiabetic therapy.

Exclusion Criteria:

* Pregnancy or lactation, use of any TZD (pioglitazone or Rosiglitazone) or insulin, renal disease or renal dysfunction , any degree of congestive heart failure, clinically significant hepatic disease or anemia, presence of unstable or severe angina or coronary insufficiency, high blood pressure

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336
Dates: Start 2000-04; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was percent change from baseline in ACR after 32 weeks of treatment. | 32 Weeks

SECONDARY OUTCOMES:
Secondary efficacy endpoints included change from baseline (visit 3) at week 32 (visit 7) in the following: serum TGF, creatinine clearance (calculated), PAI-1, CRP, IL-6, vWF, sVCAM, fibrinogen, TNF alpha, ET-1, heart rate and blood pressure | 32 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (100):
- United States (51):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Barbara, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Ukiah, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Vienna, Austria
- Canada (10):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Germany (10):
  - GSK Investigational Site, Königsfeld im Schwarzwald, Baden-Wurttemberg
  - GSK Investigational Site, Unterschneidheim, Baden-Wurttemberg
  - GSK Investigational Site, Grafing, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Borna, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Görlitz, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Apolda, Thuringia
- Latvia (4):
  - GSK Investigational Site, Jelgava
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Talsi
  - GSK Investigational Site, Valmiera
- Mexico (3):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, México
- Netherlands (4):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Zwaag
- Slovakia (3):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Martin
- Spain (5):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (7):
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Paisley, Renfrewshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Gateshead
  - GSK Investigational Site, Newport

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Bakris GL, Ruilope LM, Weston WM, Porter LE, Huang C, Heise MA, Freed MI. Rosiglitazone (RSG) added to metformin (MET) reduces urinary albumin/creatinine ratio and ambulatory blood pressure in subjects with microalbuminuria and type 2 diabetes (T2DM). Diabetes 2005;54(suppl 1):A134. Poster (543-P) presented at 65th Scientific Sessions of the Amercian Diabetes Association, June 10-14, 2005, San Diego, California.
- [Result] Ruilope LM, Bakris GL, McMorn SO, Weston WM, Huang C, Heise MA, Porter LE, Freed MI. Rosiglitazone added to metformin reduces urinary albumin/creatinine ratio and ambulatory blood pressure in subjects with microalbuminuria and type 2 diabetes. Diabetologia 2005;48(suppl 1):A283. Poster (779) presented at the 41st Annual Meeting of the European Association for the Study of Diabetes, September 12-15, 2005, Athens, Greece.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: BRL-49653/137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register